CLINICAL TRIAL: NCT05218954
Title: Posture Stability and Risk Fall Test in Objective Assessment of Balance in Patients With Ectopic Bone Tissue After Total Hip Replacement
Brief Title: Balance in Patients With Ectopic Bone Tissue After Total Hip Replacement
Status: Completed | Type: Observational
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Principal Investigator, Artur Stolarczyk, Head of the Department of Orthopedics and Rehabilitation, Medical University of Warsaw
Other Study IDs: WarsawMU/HO
Record Dates: First submitted 2022-01-19; First posted 2022-02-01 (Actual); Last update posted 2022-02-01 (Actual); Status verified 2022-01

CONDITIONS: Hip Osteoarthritis; Heterotopic Ossification; Hip Arthropathy
Keywords: total hip replacement; heterotopic ossification; hip arthritis
MeSH Terms: conditions — Osteoarthritis, Hip; Ossification, Heterotopic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients with heterotopic ossification: patients with heterotopic ossification following THR
  Interventions: Diagnostic Test: Biomechanical analysis of risk fall
- patients without heterotopic ossification: patients without heterotopic ossification following THR
  Interventions: Diagnostic Test: Biomechanical analysis of risk fall

INTERVENTIONS:
Diagnostic Test: Biomechanical analysis of risk fall — Biomechanical analysis of risk fall in terms of balance

SUMMARY:
One of the typical complications which occurs after total hip replacement (THR) procedure is heterotopic ossification (HO). According to current studies abnormal formation of bone after trauma or replacement of the hip could reach even 90% of cases. Heterotopic ossifications are causing the following symptoms, such as: pain, swelling, erythema and warmth along with joint immobility. Those factors could have an impact on maintaining the posture, especially in patients after THR.

It is well known since the 90s that the risk of fall among the population older than 65 is high. Data shows that over 30% of those people have such an incident at least once in a year. Majority of them do not have further consequences, however about 10% result in serious trauma to the head and musculoskeletal system. Falls of people who underwent THR are sometimes connected with periprosthetic fractures, which treatment is much more complicated and is associated with a higher risk of failure than treatment of ordinary fractures of the lower limb. What may even worsen the situation is that elderly people very often suffer from many diseases including osteoporosis or neoplasm which increase the risk of fracture. The rate of falls is even higher among patients hospitalised from hip fractures. In the first month after returning home about 14% of patients fall. During the 6 month period after hospitalisation it reaches 53%. So far, the influence of heterotopic ossifications on the risk of falls is unknown in the literature.

DETAILED DESCRIPTION:
This study was conducted according to the STROBE (Strengthening the Reporting of Observational studies in Epidemiology) and an appropriate checklist was presented to the editors of the Journal. Study protocol was designed as a retrospective matched-cohort observational study. This study was approved by Institutional Bioethics Committee (Number: KB/102/2007) Between January 2020 and December 2020 312 patients undergoing total hip replacement were observed. During the standard 6-weeks, 3-months and 6-months follow-up visit every patient had an AP pelvic weight-bearing x-ray. All patients were qualified and operated by a fellowship-trained single surgeon. For the present analysis, the following demographic patient data were queried: sex, age at surgery (years), and BMI. 49 patients, who developed ectopic bone formation were observed. For these patients, a propensity score based on age, sex and BMI was generated. Patients with HO were matched to patients without HO patients using a 0.1 propensity score threshold with priority given to exact matches.

All patients were operated through an anterolateral approach with the patient lying on the healthy side with one-third medium gluteal muscle dissection. Uncemented Taperloc/Allofit total hip implants (Zimmer Biomet, Warsaw, IN, USA) were used in every single case. Femoral neck dissection was performed after full joint dislocation, between the tip of the greater trochanter to the point 10 mm proximal to the lesser trochanter. Acetabular cup was placed aiming 30-40 degrees of acetabular cup inclination and 10 degrees of anteversion. Femoral stem was aimed to be placed in the anatomical axis of the femur. The postoperative protocol included chemical and mechanical thromboprophylaxis unless specifically contraindicated. All patients received one dose of parenteral antibiotics at the induction of anaesthesia and two further doses post-operatively. No pre- or postoperative ectopic bone formation prophylaxis was performed. Flexion and extension exercises of the hip, knee and ankle and isometric quadriceps contraction exercises were started on the first postoperative day, with full weight-bearing as tolerated. The aim of mobilisation with a physiotherapist was to obtain flexion of the hip of 90° mobilising and safely walking with crutches by the third postoperative day.

At 6-months follow-up visit, radiographs analysis in terms of any ectopic bone formation was performed using Brooker's classification.

All patients fulfilled WOMAC (The Western Ontario and McMaster Universities Arthritis Index) and Oxford questionnaires preoperatively and during follow-up visits.

Both cohorts underwent biomechanical assessment, performed by two independent blinded researchers (PC, KŻ) who were not aware whether patients developed ectopic bone following total hip replacement. Every analysis was performed using the Biodex Balance System (Biodex, Inc, Shirley, NY) with participants both feet standing steadily on the platform. Every participant was protected from falling with the use of support. Device screen was installed at the level of the patient's sight to avoid taking an uncomfortable position that might have influenced the results.

Postural stability test was performed, containing the results from three measurements. Every measurement has been performed on the 12th level of the platform stability for 20 seconds with 10 seconds break between every test. Results obtained from the participants were recorded as stability index (SI) values which represent deviations of platform position from the vertical in degrees. The higher SI values are, the more difficult it was for participants to maintain stability during the test.

Risk of fall test - a single test consisted of the results obtained from three measurements. Each measurement was performed at level 6 of the platform stability for 20 seconds with a 10-second rest time between attempts. The person conducting the test informed the patient in advance of how the test would proceed and then gave verbal instructions during each test. The patients were positioned in the centre of the platform, both feet set with their feet shoulder-width apart. The final result of each test was a computerised risk of fall assessment report with patient scores related to normative data.

ELIGIBILITY:
Inclusion Criteria:

* age between 60 and 80 years
* consent to particiapte in the study
* unilateral hip osteoarthritis
* primary hip osteoarthritis

Exclusion Criteria:

* neurological disorders
* diabetes mellitus
* any other surgery or lower limb injury during follow-up

Ages: 60 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients undergoing total hip replacement, who developed heterotopic ossification during 6 months postoperatively.
Sampling Method: Non-Probability Sample
Enrollment: 88 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
Postural stability test | 6 months postoperatively
  Results obtained from the participants were recorded as stability index (SI) values which represent deviations of platform position from the vertical in degrees. The higher SI values are, the more difficult it was for participants to maintain stability during the test.
Risk of fall test | 6 months postoperatively
  a single test consisted of the results obtained from three measurements. Each measurement was performed at level 6 of the platform stability for 20 seconds with a 10-second rest time between attempts. The person conducting the test informed the patient in advance of how the test would proceed and then gave verbal instructions during each test. The patients were positioned in the centre of the platform, both feet set with their feet shoulder-width apart. The final result of each test was a computerised risk of fall assessment report with patient scores related to normative data.

CONTACTS AND LOCATIONS:
Overall Officials: Artur Stolarczyk, PhD, MD, Principal Investigator — Department of Orthopedics and Rehabilitation, Medical University of Warsaw
Locations (1):
- Department of Othopedics and Rehabilitation, Medical University of Warsaw, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: Yes
IPD will be shared after rationale request from the researcher.
Supporting Information: Study Protocol